CLINICAL TRIAL: NCT01098981
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study of the Combined Lysis of Thrombus With Ultrasound and Systemic Tissue Plasminogen Activator (tPA) for Emergent Revascularization (CLOTBUST-ER) in Acute Ischemic Stroke
Brief Title: Phase 3, Randomized, Placebo-Controlled, Double-Blinded Trial of the Combined Lysis of Thrombus With Ultrasound and Systemic Tissue Plasminogen Activator (tPA) for Emergent Revascularization in Acute Ischemic Stroke
Acronym: CLOTBUST-ER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Cerevast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEREVAST THERAPEUTICS CP-01
Record Dates: First submitted 2010-04-02; First posted 2010-04-06 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Target group (Experimental): A combined treatment with transcranial US and systemic tPA
  Interventions: Device: Transcranial ultrasound as an adjunctive therapy to tPA
- Control group (Active Comparator): Systemic tPA alone
  Interventions: Drug: Standard of care tPA therapy for acute ischemic stroke

INTERVENTIONS:
Device: Transcranial ultrasound as an adjunctive therapy to tPA — * tPA per approved labeling administered over 60 minutes
  * Ultrasonic headframe with active insonation for 120 minutes
  Arms: Target group
Drug: Standard of care tPA therapy for acute ischemic stroke — * tPA per approved labeling administered over 60 minutes
  * Ultrasonic headframe with sham (inactive) insonation for 120 minutes
  Arms: Control group

SUMMARY:
This is a randomized, placebo-controlled, phase 3 clinical trial to evaluate the efficacy and safety of transcranial ultrasound (US) as an adjunctive therapy to tissue plasminogen activator (tPA) treatment in subjects with acute ischemic stroke.

DETAILED DESCRIPTION:
The primary objective of this trial is to provide information regarding the efficacy of a combined treatment with transcranial US and systemic tPA (Target group) compared to systemic tPA alone (Control group) in subjects with acute ischemic stroke. The primary efficacy endpoint is functional outcome at 3 months from stroke onset (modified Rankin Score ordinal shift analysis). The primary safety endpoint is the proportion of subjects in the Target vs Control group experiencing symptomatic intracranial hemorrhage (sICH) within 24 hours of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 - 80 years of age
2. Subjects presenting within timeframe for intravenous tPA treatment approved by local regulatory authorities but no more than 4.5 hours from onset of symptoms
3. No signs of intracranial bleeding on assessment by non-contrast CT
4. Subjects with neurological deficits of a total NIHSS score ≥ 10 points
5. Subjects that in the opinion of the treating physician require treatment with full dose IV tPA as standard of care per institutional standards
6. SBP < 185 mmHg and DBP < 105 mmHg at baseline or after treatment of hypertension with medications prior to tPA bolus
7. Pre-morbid modified Rankin score of 0-1
8. Provision of informed consent as demonstrated by the subject's signature or by the signature of the subject's authorized legal representative on the Informed Consent Form in accordance with all local and national regulations
9. Co-signature on the Informed Consent Form by a qualified member of the study staff signifying that, in his/her professional opinion, informed consent has been obtained in accordance with all local and national regulations
10. For subjects in the optional arterial recanalization substudy:

    1. Occlusion located in the intracranial carotid tee through mid M2 or proximal A2, or intracranial vertebrobasilar or P1/proximal P2 segments or tandem lesions
    2. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min for patients undergoing CTA or MRA

Exclusion Criteria:

1. Subjects with primary intra-arterial thrombolysis
2. Females who are pregnant or breast feeding
3. Subjects receiving other investigational drugs, procedures, or therapies within 30 days prior to study treatment
4. Subjects with any standard contraindication for intravenous tPA therapy
5. Significant concurrent medical/neurological conditions or test values that, in the opinion of the investigator, pose significant risk to the subject and warrant exclusion from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Modified Rankin score ordinal shift analysis | 3 months
  The primary objective of this study is to compare clinical recovery rates (modified Rankin score ordinal shift analysis) at 3 months after stroke onset.

SECONDARY OUTCOMES:
Symptomatic intracerebral hemorrhage | 0-24 hours from treatment
  The secondary outcome is a comparison of the rates of symptomatic intracerebral hemorrhage within 0-24 hours from initiation of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cerevast Therapeutics, Inc., Redmond, Washington, United States

REFERENCES:
- [Derived] Alexandrov AV, Kohrmann M, Soinne L, Tsivgoulis G, Barreto AD, Demchuk AM, Sharma VK, Mikulik R, Muir KW, Brandt G, Alleman J, Grotta JC, Levi CR, Molina CA, Saqqur M, Mavridis D, Psaltopoulou T, Vosko M, Fiebach JB, Mandava P, Kent TA, Alexandrov AW, Schellinger PD; CLOTBUST-ER Trial Investigators. Safety and efficacy of sonothrombolysis for acute ischaemic stroke: a multicentre, double-blind, phase 3, randomised controlled trial. Lancet Neurol. 2019 Apr;18(4):338-347. doi: 10.1016/S1474-4422(19)30026-2. PMID 30878103
- [Derived] Schellinger PD, Alexandrov AV, Barreto AD, Demchuk AM, Tsivgoulis G, Kohrmann M, Alleman J, Howard V, Howard G, Alexandrov AW, Brandt G, Molina CA; CLOTBUSTER Investigators. Combined lysis of thrombus with ultrasound and systemic tissue plasminogen activator for emergent revascularization in acute ischemic stroke (CLOTBUST-ER): design and methodology of a multinational phase 3 trial. Int J Stroke. 2015 Oct;10(7):1141-8. doi: 10.1111/ijs.12536. Epub 2015 Jun 29. PMID 26120902